CLINICAL TRIAL: NCT02674139
Title: Comparative Study of Intrauterine Contraceptive Device Insertion During Caesarean Section Versus Conventional Application
Brief Title: Comparison Between Intrauterine Contraceptive Device Insertion During Cesarean Section Vs Conventional Application
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: sara AbdAllah (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Sponsor-Investigator, sara AbdAllah, Assistant lecturer of Obstetrics and Gynecology Faculty of Medicine- Beni-sueif University, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO-MD-IUD
Record Dates: First submitted 2016-01-30; First posted 2016-02-04 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Contraception
Keywords: post placental-caesarean-IUD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IUD insertion 6 Weeks after delivery (Active Comparator): Subjects randomized to interval placement will have their Copper T 380A IUD placed in the office at six weeks postpartum or later
  Interventions: Device: Copper T 380A IUD
- Immediate Post-placental insertion (Experimental): Subjects randomized to receive the Copper T 380A IUD within 10 minutes of delivery of the placenta during caesarean section.
  Interventions: Device: Copper T 380A IUD

INTERVENTIONS:
Device: Copper T 380A IUD — intrauterine contraceptive device T-shaped loaded with cupper
  Other Names: Pregna

SUMMARY:
The study aims to compare immediate post-placental (within 10 minutes of placenta delivery) intrauterine contraceptive device (Copper T 380A) insertion versus conventional placement at 6 weeks (often referred to as delayed or interval insertion) regarding the clinical outcomes (safety, efficacy, expulsion and continuation rates) for women undergoing caesarean section.

DETAILED DESCRIPTION:
• Study Design: A controlled randomized clinical trial (CRCT)

• Study Site: The study will be carried out in the Department of Obstetrics and Gynecology at Beni-suef University Hospital

• Study Population: The study population will include pregnant women between 36-40 weeks gestational ages who attend antenatal care and are eligible for insertion of IUCD during delivery through elective caesarean section.

• Study Sample: The study will consist of 200 women which will be chosen randomly to whom elective lower segment caesarean section will be done at the Obstetrics and Gynecology department, willing to have an intrauterine device (IUD) inserted for postpartum contraception and willing to comply with the study protocol.

After informed consent is obtained, eligible study participants will be randomized into 2 groups:

Group (A): 100 Women will receive the Pregna ® IUD at the 6 week postpartum visit Group (B): 100 Women will receive the Pregna ® IUD within 10 minutes of delivery of the placenta during caesarean section.

• Study Procedure:

Insertion Technique:

During caesarean section:

Uterine cavity will be inspected for presence of malformations following placental delivery, which would limit use of IUCD.The IUCD (Pregna Copper T 380A) will be removed from the insertion sleeve and will be placed on the sterile field. Uterus is stabilized by grasping it at fundus. Insertion will be done during cesarean delivery, after ex pulsion of placenta and through the uterine incision, manually (IUCD is Held between middle and index finger). It will be inserted into the uterus through uterine incision and will be released at fundus of uterus. Hand will be removed slowly from the uterus. Enough care will be taken not to dislodge IUCD as hand is removed. Strings will be guided toward the lower uterine segment without disturbing IUCD'S fundal position. Enough Care will be taken not to include IUCD strings during uterine closure.

Delayed postpartum IUDs Will be inserted in the usual sterile fashion as described in the manufacturer's instructions at the 6-week postpartum visit

Later Prior to Discharge:

* IUCD Client card, showing type of IUCD and date of insertion will be given to patient.
* She will be informed about the IUCD side effects and normal postpartum symptoms.

  * Patients will be scheduled for a control examination at 1 week, 6 weeks, 3 months and 6 months after the insertion.
  * She will be advised to contact one of the physicians immediately if they experienced:-
  * Unusual vaginal discharge different from the usual lochia.
  * Lower abdominal pain, especially if accompanied by fever or chills.
  * Feeling of being pregnant.
  * Suspicion that the IUCD has fallen out.

Follow up visits:

* At each visit the patients will be questioned for symptoms of expulsion, excessive bleeding and infection. In addition, a pelvic examination (per speculum) and trans-vaginal ultrasound will be performed at each follow-up visit.
* In per speculum examination if IUD threads are long, they will be cut 2 cm from external os. If threads of IUD are not seen and there was no history of expulsion of IUD, pelvic ultrasonography or X-ray pelvis will be done to note for misplaced IUD.
* All the patients will subjected to the follow up:
* The IUD will be removed in the case of partial expulsion, bleeding or pain, or at the patient's request.

  * Ethical Considerations

    1-Approval by the institution ethical committee 2-Individual Consent Process: Written informed consent will be taken after explaining the study objective the procedures to potential participants. Participation will be voluntary and participants will be informed that the decision not to participate will not impact on the quality of care they receive.
  * The statistical Analysis:

Data will be statistically described in terms of mean + standard deviation (+/- SD), frequencies (number of cases) and relative frequencies (percentages) when appropriate. Comparison of numerical variables between the study groups will be done using Student t test for independent samples. For comparing categorical data, Chi square (X2) test will be performed. Exact test will be used instead when the expected frequency is less than 5. P values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Age: 18 - 45 years.
* GA 36-40 weeks based upon the date of last normal menstruation, confirmed by ultrasonographic scan.
* Desire to have intrauterine contraceptive device (Cu T) after counseling about different contraceptive options and consented to the study.

Exclusion criteria:

* Allergy to copper.
* Ante- or intra-partum hemorrhage.
* Hemorrhagic disorders.
* Current or past history of pelvic inflammatory disease.
* Women known to have pelvic TB.
* Known to have ruptured membranes for more than 24 h prior to delivery.
* History of chorioamnionitis.
* Known uterine abnormalities e.g., Bicornuate/septate Uterus, uterine myoma.
* Patients presented with febrile morbidity prior to the operation defined as temperature above 38'c.
* Multiple pregnancies.
* Placenta previa.
* History of ectopic pregnancy.
* Anemia (hemoglobin <10 g/dl).
* Cervical cancer or carcinoma in situ.
* Diagnosis of active cervical infection for standard insertion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Expulsion: Complete IUD expulsion will be verified clinically and by transvaginal ultrasound | 6 months
  Complete IUD expulsion will be verified clinically and by transvaginal ultrasound. An IUD will be considered to be partially expelled if a distance greater than 10 mm is measured between the vertical arm of the IUD and the junction between the endometrium and the uterine cavity)

SECONDARY OUTCOMES:
Uterine perforation (assessed by pelvic ultrasonography or X-ray) | 6 months
  To be assessed by pelvic ultrasonography or X-ray pelvis will to note for misplaced IUD
Pelvic pain (using the 0-10 Numeric Pain Rating Scale) | 6 months
  Using the 0-10 Numeric Pain Rating Scale and analgesic doses required
Strings not visible (assessed by speculum examination) | 6 months
  To be assessed by speculum examination.
Pelvic infection: number of participants with Pelvic infection | 6 months
  number of participants with Pelvic infection
Psychological (satisfied or not) using questionnaire | 6 months
  using questionnaire
Pregnancy (assessed by serum pregnancy test and pelvic ultrasound) | 6 months
  To be assessed by serum pregnancy test and pelvic ultrasound in suspicious cases (missed period - misplaced IUD - expelled IUCD either partial or complete)

CONTACTS AND LOCATIONS:
Overall Officials: sara AA mohamed, master, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided